CLINICAL TRIAL: NCT06847243
Title: Effect of Nutrigenetic Intervention on Cardiovascular Biomarkers, Oxidative Stress and Antioxidant Capacity in Subjects with Abdominal Obesity
Brief Title: INNUPREC (Nutrigenetic Intervention for the Prevention of Cardiovascular Disease)
Acronym: INNUPREC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, ERIKA MARTINEZ-LOPEZ, Principal Investigator, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CI-05223
Record Dates: First submitted 2025-02-10; First posted 2025-02-26 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Abdominal Obesity
Keywords: Abdominal obesity; Nutrigenetic intervention; Cardiometabolic biomarkers
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Intervention Model Description: Randomized parallel clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutrigenetic intervention (Active Comparator)
  Interventions: Diagnostic Test: Nutrigenetic diet according the genetic test
- Control Intervention (Placebo Comparator)
  Interventions: Other: Control intervention group

INTERVENTIONS:
Diagnostic Test: Nutrigenetic diet according the genetic test — Subjects within the nutrigenetic intervention group will be provided with a dietary plan according to nutrient intake characteristics by alghoritm genetic afinity.
  Arms: Nutrigenetic intervention
Other: Control intervention group — Subjects within the control intervention group will be provided with a dietary plan according to general nutrient recommendation by the AHA (American Hearth association) and national cholesterol education program
  Arms: Control Intervention

SUMMARY:
Background: Abdominal obesity (AO) is a multifactorial disease that affects 81.6% of the Mexican population; it is characterized by the excessive accumulation of adipose tissue in abdominal region. Scientific evidence suggest that regional fat distribution plays a critical role in the development of cardiovascular diseases (CVD). The main processes involved in the increased risk of developing CVD in the presence of AO are alterations in insulin signaling, dyslipidemias, atherosclerosis, inflammation, and oxidative damage. On the last years has been reported genetic variations associated with AO and dyslipidemia. In addition, interactions have been found between these genetic variants and diet that may be influencing a differential response in metabolic, molecular, and phenotypic processes, which favor the development of CVD. Objective: Evaluate the effect of nutrigenetic intervention on cardiovascular biomarkers, oxidative stress and antioxidant capacity in subjects with abdominal obesity. Materials and methods: The present study is a simple randomized clinical trial. Participants will be randomized into one of two groups of intervention; Control group and Nutrigenetic group during a 2-month follow-up period. Anthropometric, dietary evaluation and biochemical markers assessments will be monitored at baseline, at 4 weeks (mid-intervention), and at 8 weeks (end of intervention). The dietary evaluation was analyzed by Nutritionist Pro software. Body composition was evaluated by electrical bioimpedance (InBody 370). All biochemical determinations were analyzed by dry chemistry (Vitros 350) and cardiometabolic markers by colorimetric immunoassay technology. Infrastructure: Institute of Translational Nutrigenomics and Nutrigenomics, University Center for Health Sciences, University of Guadalajara.

DETAILED DESCRIPTION:
A total of 60 subjects will be invited to enroll in a clinical trial of nutrigenetic or control intervention. Prior to randomization and the start of the intervention, all subjects will be scheduled for a first appointment where their medical history will be taken and a blood sample will be taken for DNA extraction and their genetic profile will be performed (including 21 SNV (single nucleotide variation) involved in cardiometabolic disorders). The assignment to the intervention group will be done through a random permuted block assignment. In the case of the subjects of the nutrigenetic intervention group, with the help of an algorithm designed for the purposes of this study, their genetic profile of the variants of interest will be entered, in order to determine the dietary pattern to which they have the greatest affinity. Once this data is available, they will be given their eating plan. Regarding the control group, the characteristics of their menu will adhere to what is established in a correct diet and the recommendations of the American Heart Association.

This clinical trial will consist in a 8-week intervention with recurrent visits every 4 weeks. Subjects will be required to follow the dietary plan provided in a menu produced and edited by our research group. In every visit, all subjects will undergo a body composition analysis as well as blood tests that include: total cell count, glucose and lipid homeostasis, serum oxidative and antioxidant markers. In total, they will be evaluated anthropometrically and biochemically on 3 occasions, at baseline, 1 month and 2 months (final).

This study proposes three distinct but closely related approaches to gain a better understanding of nutrigenetics and its impact on precision nutrition.

* To compare the effect and impact of personalized nutritional interventions on nutritional diets with general recommendations.
* See the impact of a personalized diet in improving parameters involved in the development of cardiovascular diseases
* Develop new personalized nutritional treatment strategies for subjects with chronic diseases

Once the project is finished, new research strategies will be proposed for future studies, seeking to have an evaluation beyond the anthropometric and biochemical, such as microbiota or gene regulation. In addition to this, the application of the knowledge generated in the project to the health care of patients with obesity who may come to our service in the future will be encouraged. Finally, the knowledge generated will be disseminated in our institutional community, which would increase the impact and significance of the project.

In summary, the impact of this study is divided into the following points:

* Design of new strategys as nutrigenetic intervention´s for the treatment and prevention metabolic disease such as obesity and cardiovascular
* Identification of some cardiovascular biomarkers relevant to the treatment of abdominal obesity and its comorbidities
* Useful information on gene-nutrient interaction for the public and private sector in the field of genetic testing
* Study population benefited from the results of the intervention and the information of their genetic and biochemical profiles

ELIGIBILITY:
Inclusion Criteria:

* 30-65 years of age
* Subjects who agree to participate in the study and all signed informed consent
* Women with a waist circumference ≥ 88 cm and men ≥ 102 cm according to NCEP/ATPIII.

Exclusion Criteria:

* Currently consuming any of the following drugs: NSAIDs, anticoagulants, hypoglycemic, or hypolipemic drugs
* Diagnosed autoimmune diseases
* Diagnosed cancer
* Pregnancy and breastfeeding
* Subjects who have undergone a dietary intervention at the time or up to 3 months prior
* Subjects who wish to abandon the study

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Waist Circumference between nutrigenetic and control group | At baseline, first month and second month (final)
  Waist circumference is used as a diagnostic criterion for abdominal obesity, which is why it is the main change to be evaluated among our study groups.
  Waist circumference will be measure at the narrowest point between the edge of the inner rib and the iliac crest, with the participant in an abducted and relaxed position, after expiration using a Lufkin Executive® tape.

SECONDARY OUTCOMES:
Changes in Weight | At the baseline (0 Month) and 1st month, 2nd month (final)
  The weight will be measure in kilograms on InBody 370
Changes in Fat Mass | At the baseline (0 Month) and 1st month, 2nd month (final)
  The Fat Mass will be measure in kilograms by electrical bioimpedance on InBody 370
Changes in Total Cholesterol | At the baseline (0 Month) and 1st month, 2nd month (final)
  Will be measure in mg/dL using a dry chemistry system in Vitros 350 equipment.
Changes in Triglycerides | At the baseline (0 Month) and 1st month, 2nd month (final)
  Will be measure in mg/dL using a dry chemistry system in Vitros 350 equipment.
Changes in High-density lipoprotein (c-HDL) | At the baseline (0 Month) and 1st month, 2nd month (final)
  Will be measure in mg/dL using a dry chemistry system in Vitros 350 equipment.
Changes in Low-density lipoprotein (c-LDL) | At the baseline (0 Month) and 1st month, 2nd month (final)
  Will be calculated using Friedewald formula, which uses the parameters of total cholesterol, HDL and VLDL and the result is reported in mg/dL
Changes in serum glucose | At the baseline (0 Month) and 1st month, 2nd month (final)
  Will be measure in mg/dL using a dry chemistry system in Vitros 350 equipment.
Changes in serum insulin | At the baseline (0 Month) and 1st month, 2nd month (final)
  It be measure by chemiluminescence immunoassay in DiaSorin Liaison equipment
Changes in homeostatic model assessment - insulin resistance (HOMA-IR) | At the baseline (0 Month) and 1st month, 2nd month (final)
  Serum glucose and Insulin levels were be combined to report HOMA-IR calculated as described by Matthews
Changes in serum Oxidized low-density lipoprotein (oxLDL) | At the baseline (0 Month) and 1st month, 2nd month (final)
  Will be measured in pg/dL. Serum oxLDL levels will be quantified according to the supplier's instructions by an enzyme linked immunosorbent assay (ELISA) kit provided by Cell Biolabs, Inc
Changes in serum Oxidized high-density lipoprotein (oxHDL) | At the baseline (0 Month) and 1st month, 2nd month (final)
  Will be measured in pg/dL. Serum oxHDL levels will be quantified according to the supplier's instructions by an enzyme linked immunosorbent assay (ELISA) kit provided by Cell Biolabs, Inc
Changes in serum Total antioxidant capacity | At the baseline (0 Month) and 1st month, 2nd month (final)
  Will be measure from serum samples using an OxiSelect TAC Assay Kit, (Cell Biolabs) and reported in mM.
Changes in serum Lipid peroxidation | At the baseline (0 Month) and 1st month, 2nd month (final)
  Will be measure in μM. Serum lipid peroxidation will be quantified according to the supplier's instructions by Lipid peroxidation assay kit, Oxford Biomedical
Changes in hsPCR | At the baseline (0 Month) and 1st month, 2nd month (final)
  Serum levels will be measure using an automated biochemical analyzer, Mindray BS-120 chemistry analyzer, from Shenzhen Mindray Bio-Medical Electronics Co.
Changes in ApoA1 | At the baseline (0 Month) and 1st month, 2nd month (final)
  Serum levels will be measure using an automated biochemical analyzer, Mindray BS-120 chemistry analyzer, from Shenzhen Mindray Bio-Medical Electronics Co.
Changes in ApoB | At the baseline (0 Month) and 1st month, 2nd month (final)
  Serum levels will be measure using an automated biochemical analyzer, Mindray BS-120 chemistry analyzer, from Shenzhen Mindray Bio-Medical Electronics Co.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Campos-Perez, PhD, Study Chair — University of Guadalajara; Alondra Mora-Jiménez, Graduate, Study Chair — University of Guadalajara
Locations (1):
- University of Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared to protect and safeguard the confidentiality data of the participants.